CLINICAL TRIAL: NCT05342662
Title: Evaluating the Consequences of Mistimed Light-emitting Device Use on Cardiac Activity and Sleep Health
Brief Title: Light Sleep: Screen Use and Sleep Health
Acronym: LS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Responsible Party: Principal Investigator, David Reichenberger, Principal Investigator, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: STUDY00019746
Record Dates: First submitted 2022-04-06; First posted 2022-04-25 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Glasses
MeSH Terms: interventions — Eyeglasses

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to wear either blue light-blocking glasses or glasses with clear lenses during the second week of the study. During the third week, participants will be assigned to wear the opposite pair of glasses. Sleep and wake behaviors are the primary study outcome.
Who Masked: Participant
Masking Description: Participants will be told that both pairs of glasses block blue light.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blue light-blocking glasses (Experimental): Participants will wear blue light-blocking glasses to evaluate whether sleep behaviors improve.
  Interventions: Device: Blue light-blocking glasses
- Glasses with clear lenses (Placebo Comparator): Participants will wear glasses with clear lenses to serve as the control condition.
  Interventions: Device: Glasses with clear lenses

INTERVENTIONS:
Device: Blue light-blocking glasses — Participants will be randomly assigned to wear either blue light-blocking glasses or glasses with clear lenses during the second week of the study. During the third week, participants will be assigned to wear the opposite pair of glasses.
  Other Names: Swanwick Night Swannies
  Arms: Blue light-blocking glasses
Device: Glasses with clear lenses — Non-blue light-blocking glasses
  Other Names: Swanwick glasses
  Arms: Glasses with clear lenses

SUMMARY:
The Phone Sleep Study is being done to find out whether wearing blue light-blocking glasses in the evening improves subsequent sleep. This is a 21-day study and participants will be asked to wear a sleep-monitoring "actiwatch", a heart tracker, and an activity monitor, as well as to provide screenshots of participants' smartphone's screen time app for three weeks. Participants will also be asked to wear a blood pressure cuff on their arm for three days during each week, for a total of nine days.

ELIGIBILITY:
Inclusion Criteria:

1. Fluent English speaker and reader
2. Capable of providing one's own informed consent
3. Age 18 to 29 years old
4. Healthy, sighted individuals
5. Own an iOS smartphone (iPhone)
6. Willingness to update smartphone to access the current version of the Screen Time or StayFree application, depending on smartphone operating system
7. Willingness to participate in surveys, wear health monitoring devices, and provide screenshots of their smartphone's screentime application throughout the entire study

Exclusion Criteria:

1. Younger than 18 or older than 29 years
2. Individuals who are blind or wear corrective lenses
3. Taking prescribed medications that affect sleep
4. Recent shift work
5. Sleep disorder diagnosis or any cardiovascular disease

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2022-11-23 (Actual); Primary Completion 2023-09-05 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Sleep onset | Throughout the duration of the study (~3 weeks)
  Midnight-centered clocktime of when participant falls asleep at night
Sleep midpoint | Throughout the duration of the study (~3 weeks)
  Midnight-centered clocktime denoting the middle of the nocturnal sleep episode
Total sleep time at night | Throughout the duration of the study (~3 weeks)
  Length of time spent asleep during the night, excluding time spent awake throughout the sleep episode

CONTACTS AND LOCATIONS:
Overall Officials: David Reichenberger, MS, Principal Investigator — Department of Biobehavioral Health
Locations (1):
- Biobehavioral Health Building, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
All processed IPD data that underlie results in a publication
Supporting Information: Analytic Code
Time Frame: Starting 1 year after the last publication based on collected data
Access Criteria: Interested parties should contact David Reichenberger (reichenberger@psu.edu)